CLINICAL TRIAL: NCT07407426
Title: Effects of EEG-guided Binaural Beat Audio Intervention on Brain Reactivity Associated With Performance-related Stress and Cognition Among Professional Musicians: A Randomized, Double-blinded, Sham-controlled Functional Neuroimaging Trial
Brief Title: EEG-Guided Binaural Beat Audio to Reduce Performance-Related Stress and Improve Cognition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: Texas Tech University (Other)
Responsible Party: Principal Investigator, Samudani Dhanasekara, Assistant Professor, Texas Tech University Health Sciences Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB2025-681
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Cognitive Abilities; Performance; Stress; Cognitive Performance
Keywords: neurofeedback; cognitive performance; stress

STUDY DESIGN:
Masking Description: Double (Participant, Outcomes Assessor/Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EEG-guided binaural beat audio (Experimental): 30-minute session delivered via headphones; proprietary algorithm uses real-time single-electrode EEG from the left prefrontal cortex to dynamically adjust binaural beat frequencies.
  Interventions: Other: EEG-guided binaural beat audio
- non-binaural audio (Sham Comparator): 30-minute session of music without frequency differences between ears (non-binaural), delivered via identical headphones; blinding maintained.
  Interventions: Other: Non-binaural audio intervention

INTERVENTIONS:
Other: EEG-guided binaural beat audio — 30-minute session delivered via headphones; proprietary algorithm uses real-time single-electrode EEG from the left prefrontal cortex to dynamically adjust binaural beat frequencies.
  Arms: EEG-guided binaural beat audio
Other: Non-binaural audio intervention — 30-minute session of music without frequency differences between ears (non-binaural), delivered via identical headphones; blinding maintained.
  Arms: non-binaural audio

SUMMARY:
Performance-related stress can impair sustained attention, inhibitory control, and memory. This randomized, double-blinded, sham-controlled parallel-arm trial evaluates whether a 30-minute EEG-guided binaural beat audio intervention reduces subjective stress/performance anxiety and improves cognition, and whether it changes task-related brain reactivity measured by fMRI. The intervention uses real-time single-electrode EEG recorded over the left prefrontal cortex to dynamically adjust binaural beat frequencies to guide the brain toward a target state; the sham condition uses non-binaural music delivered through identical headphones.

Adult music majors preparing for an upcoming concert will complete pre- and post-intervention fMRI sessions during cognitive/music tasks (Stop Signal Reaction Task, Music Reading Task, Music Memory Retrieval Task) and complete visual analog scales (VAS) assessing performance anxiety, stress, and related subjective states. The primary outcomes include fMRI task-related activity in stress-regulation regions (dlPFC, amygdala, hippocampus), behavioral inhibition indices from the stop-signal task, music memory retrieval accuracy, and VAS-reported stress/performance anxiety.

DETAILED DESCRIPTION:
This study will test the efficacy and neurophysiologic mechanism of a novel EEG-guided binaural beat audio intervention for mitigating performance-related stress and enhancing cognition in musicians. The study is conducted at Texas Tech University (recruitment/screening/analysis) with neuroimaging and cognitive task data collection at the Texas Tech Neuroimaging Institute (TTNI).

Participants complete a single in-person visit (~3 hours) including consent and eligibility screening, task training, pre-intervention VAS and fMRI scanning, randomization to intervention or sham, a 30-minute audio session, post-intervention fMRI scanning, and post-intervention VAS.

The experimental audio intervention uses a proprietary algorithm with real-time EEG feedback from a single electrode over the left prefrontal cortex to dynamically adjust binaural beat frequencies during a 30-minute session delivered through headphones. The sham comparator uses non-binaural audio (music without interaural frequency differences) delivered identically. Participants and researchers conducting assessments are blinded to allocation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+ years) enrolled as undergraduate music majors at Texas Tech University
* Currently preparing for an upcoming concert performance within the next 3 months
* Able to read standard musical notation

Exclusion Criteria:

* Subjects with contraindications to undergo MRI after being screened by the TTNI safety screening sheet - specifically, Subjects with implanted devices that are not compatible with MRI including, but not limited to cardiac pacemakers, cardiac defibrillators, aneurysm clips, carotid artery vascular clamps, implanted nerve stimulators (neuron-stimulators also called TENS or wires), bone growth or bone fusion stimulators, cochlear implants, vagus nerve stimulators, filters for blood clots (Umbrella, Greenfield, bird's nest), embolization coils (e.g. Gianturco) in the brain, ocular implants, vascular stents, medication pumps, medication patches delivering medications, implanted limbs, ventricular shunts, metal joints, rods, plates, pins, screws, nails, or clips, penile implants, or contraceptives devices including IUDs, cervical pessaries and diaphragms Subjects who have undergone cataract surgery Subjects who have shrapnel or metal in the head, eyes or skin Subjects with a history of working with metal fragments ( or have had metal removed from eyes Subjects with gunshot wounds or BB gun injury Subjects with permanent metal body piercings or jewelry that cannot be removed Subjects who use hearing aids or have braces / permanent retainers that cannot be removed temporarily for the MRI scans Subjects with large tattoos in the head and neck area Subjects with claustrophobia Subjects who are currently pregnant or suspected to be pregnant
* Physical, medical, neurological or psychiatric impairments (including substance abuse)
* Current use of medications that could affect cognitive performance (including beta-blockers, stimulants, anxiolytics, antidepressants, or antipsychotics)
* History of head injury resulting in loss of consciousness/history of brain surgery
* History of diagnosed hearing impairment or use of hearing aids
* Current or past diagnosis of epilepsy or seizure disorders
* Unwillingness or inability to refrain from alcohol consumption 48 hours prior to the study visit
* Unwillingness or inability to refrain from caffeine consumption 12 hours prior to the study visit
* Current/past history of substance abuse
* Pregnancy or possibility of pregnancy
* Unwillingness or inability to follow written, on-screen, and verbal instructions given by the study team

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
fMRI task-related activity | Baseline (immediately prior to 30-minute intervention/control audio session) and immediately post-intervention/control audio session (within 30 minutes after completion of session).
  fMRI task-related activity in dlPFC, amygdala, hippocampus during SSRT, MRT, MMRT (see below).

SECONDARY OUTCOMES:
Stop Signal Reaction Time | Baseline (immediately prior to 30-minute intervention/control audio session) and immediately post-intervention/control audio session (within 30 minutes after completion of session).
  Estimated time (milliseconds) required to inhibit a prepotent response following a stop signal, computed using the horse-race model and drift-diffusion theory. Lower values indicate better inhibitory control.
Music Reading Task | Baseline (immediately prior to 30-minute intervention/control audio session) and immediately post-intervention/control audio session (within 30 minutes after completion of session).
  Subjects will be presented with images of musical staffs and asked to read the music in their minds, as if they were playing their instrument during the concert. Forty out of 80 images will be taken from the subject's own concert repertoire. Twenty other images will be taken from the subject's concert, with alterations, and another 20 from their classmates' concerts. The activation of mirror neurons will be detected by fMRI. fMRI reactivity of especially mirror neuron-related regions, in addition to the brain regions noted above under the fMRI section will be examined during the task as the main outcome of the task.
Music Memory Retrieval Task | Baseline (immediately prior to 30-minute intervention/control audio session) and immediately post-intervention/control audio session (within 30 minutes after completion of session).
  Subjects will be presented with images of staff. They will answer whether they saw the staff during the previous task using a hand-held device with designated response buttons. Proportion of images correctly identified as "seen." Range 0-1; higher values indicate better recognition sensitivity. The unit of measurement is in proportion (0-1) assigned as the hit rate.
Visual Analogue Scale - Stress | Baseline (immediately prior to 30-minute intervention/control audio session) and immediately post-intervention/control audio session (within 40 minutes after completion of session).
  100 mm VAS, anchored at 0 ("Not Stressed") and 100 ("Stressed"). Higher scores = greater stress.
Visual Analogue Scale - Confidence of Performance | Baseline (immediately prior to 30-minute intervention/control audio session) and immediately post-intervention/control audio session (within 40 minutes after completion of session).
  100 mm VAS, anchored at 0 ("Not confident at all") and 100 ("Extremely confident"). Higher scores = greater perceived confidence in performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data may be shared with qualified researchers upon a reasonable request and after obtaining institutional approval, as the study is based on a proprietary algorithm owned by Texas Tech University.